CLINICAL TRIAL: NCT03913702
Title: Subacromial Injection of Methylprednisolone Versus Ketorolac to Treat Shoulder Impingement: a Double-blind Randomized Controlled Trial
Brief Title: Subacromial Methylprednisolone Versus Ketorolac for Shoulder Impingement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate patient enrollment
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTMB IRB #: 18-0156
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Subacromial Impingement; Subacromial Impingement Syndrome
Keywords: Ketorolac; Methylprednisolone; Subacromial impingement syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Ketorolac Tromethamine; Methylprednisolone Acetate

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial in which patients will be randomized to receive subacromial injection with either methylprednisolone or ketorolac.
Who Masked: Participant, Investigator
Masking Description: Neither the treating physician nor the patient will have access to drug-related details. Data will only be retrieved by the coordinating institution's research coordinator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac (Active Comparator): Assigned patients will receive a subacromial injection of ketorolac 60mg (2ml + 8ml lidocaine 1%)
  Interventions: Drug: Ketorolac Tromethamine
- Methylprednisolone (Active Comparator): Assigned patients will receive a subacromial injection of methylprednisolone 80mg (1ml + 9ml lidocaine 1%)
  Interventions: Drug: Methylprednisolone Acetate

INTERVENTIONS:
Drug: Ketorolac Tromethamine — 2ml of injectable Ketorolac (30mg/ml) will be mixed with 8ml of lidocaine HCL (1% without epinephrine) and delivered into the subacromial joint (total of 60mg of active substance in 10ml).
  Other Names: Toradol
  Arms: Ketorolac
Drug: Methylprednisolone Acetate — 1ml of injectable Methylprednisolone (80mg/ml) will be mixed with 9ml of lidocaine HCL (1% without epinephrine) and delivered into the subacromial joint (total of 80mg of active substance in 10ml)
  Other Names: DepoMedrol
  Arms: Methylprednisolone

SUMMARY:
The investigators aim to compare subacromial ketorolac (non-steroidal anti-inflammatory drug) versus methylprednisolone (steroid) for the treatment of shoulder impingement syndrome.

DETAILED DESCRIPTION:
Because of the current conflicting evidence, the lack of long-term follow-up, and the multiple potential benefit benefits to the society, the investigators aim to compare subacromial ketorolac versus methylprednisolone for the treatment of shoulder impingement syndrome. The investigators hypothesize that patients with shoulder impingement treated with a subacromial methylprednisolone versus ketorolac have similar outcomes based on the ASES (American Shoulder and Elbow Surgeon) self-assessment score. The study will be performed at one institution, the University of Texas Medical Branch.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Severe or recalcitrant shoulder impingement syndrome
* Subacromial injection is a therapeutic option

Exclusion Criteria:

* Allergy or intolerance to steroids within less than 1 month
* Allergy or intolerance to NSAIDs within less than 1 month
* Pregnancy
* Breastfeeding
* Pre-existing asthma
* Uncontrolled psychiatric illness
* Previous shoulder injection within the past 3 months
* Evidence of confounding shoulder pathology on imaging
* History of a full-thickness rotator cuff tear
* Ipsilateral cervical radiculopathy
* Moderate to severe glenohumeral arthritis
* Systemic inflammatory conditions
* Kidney disease
* Liver disease
* Gastrointestinal ulcer
* Bleeding disorder
* Pending litigation or work-related claims related to the shoulder
* Previous shoulder surgery on the affected shoulder
* Evidence of local infection
* Evidence of adhesive capsulitis
* Evidence of shoulder instability

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Somerson, MD, Principal Investigator — University of Texas
Locations (1):
- Universtiy of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
At the end of this investigation, IPD-related results will be tabulated and submitted to clinicaltrials.gov to report. This would help evaluate the effects and safety of interventions administered.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 20 weeks from the last patient enrollment
Access Criteria: At the end of this investigation, all results will be tabulated and submitted to clinicaltrials.gov to report.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Early termination due to inadequate patient enrollment.
Period: Overall Study
Arm/Group | Ketorolac | Methylprednisolone
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant enrolled in the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Methylprednisolone | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Surgeon (ASES)
Description: The ASES is a self-assessment score, ranging between 0 and 100 (0 indicating the worst shoulder condition and 100 indicating the best shoulder condition), applicable for use in patients with shoulder pathology. A higher pain score indicates the subject is in more pain. A lower pain score indicates less pain.
Time Frame: 12 weeks
Population: No data collected.
Arm/Group | Ketorolac | Methylprednisolone
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: American Shoulder and Elbow Surgeon (ASES)
Description: as for outcome 1
Time Frame: 2 weeks
Population: No data collected.
Arm/Group | Ketorolac | Methylprednisolone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: American Shoulder and Elbow Surgeon (ASES)
Description: The ASES is a self-assessment score, ranging between 0 and 100, (0 indicating the worst shoulder condition and 100 indicating the best shoulder condition), applicable for use in patients with shoulder pathology. A higher pain score indicates the subject is in more pain. A lower pain score indicates less pain.
Time Frame: 4 weeks
Population: No data collected.
Arm/Group | Ketorolac | Methylprednisolone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Range of Motion (ROM)
Description: The range of motion is a function-related measure, that reflects the extent of shoulder movement (measured in degrees, in forward flexion, and abduction with internal/external rotation of the shoulder)
Time Frame: 12 weeks
Population: No data collected.
Arm/Group | Ketorolac | Methylprednisolone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Description: The protocol was discontinued early.
Arm/Group | Ketorolac | Methylprednisolone
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
The protocol was terminated early due inadequate patient enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT03913702/Prot_SAP_001.pdf